CLINICAL TRIAL: NCT04105595
Title: Multi Centre, International, Post Market Registry to Monitor the Clinical Performance and Safety of an Atrial Septal Closure Device With Bioresorbable Framework in Patients With Clinically Significant Atrial Septum Defect (ASD) or Patent Foramen Ovale (PFO) in Routine Clinical Use
Brief Title: Post Market Registry of the CBSO
Acronym: CBSO Registry
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: atHeart Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: 2019.8408
Record Dates: First submitted 2019-09-24; First posted 2019-09-26 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Atrial Septal Defect; Patent Foramen Ovale
MeSH Terms: conditions — Heart Septal Defects, Atrial; Foramen Ovale, Patent

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ASD patients
  Interventions: Device: Septal defect closure
- PFO patients
  Interventions: Device: Septal defect closure

INTERVENTIONS:
Device: Septal defect closure — Device closure of atrial septal defect

SUMMARY:
Multi centre, international, post market registry to monitor the clinical performance and safety of an atrial septal closure device with biodegradable framework in patients with clinically significant atrial septum defect (ASD) or patent foramen ovale (PFO) in routine clinical use

ELIGIBILITY:
Inclusion Criteria:

* Patient suffers from ASD (including ostium secundum ASD or a fenestration from a Fontan procedure) or PFO and is planned to receive the CBSO.
* Patient (or legal guardian) has been informed and agreed to and signed the informed consent form.
* A CBSO is implanted into the patient.

Exclusion Criteria:

* Patient is known to have one or more of the contraindications listed in the instructions for use.
* Patient is currently participating in one or more interventional studies, with exception of a study investigating the CBSO.
* Patient is implanted with another product in the atrial septum.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Intent to treat population: All enrolled patients Modified Intent to Treat population: All enrolled patients who have a permanently implanted CBSO.
  Per Protocol population: All patients in the enrolled population who have a permanently implanted CBSO and do not have a major protocol deviation. The per protocol population will be used as the final population for analysis.
Sampling Method: Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2020-03-05 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Effective closure by echocardiography | at 6 months
Safety throughout the follow up duration by absence of serious incidents | day 0 to 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Deutsches Herzzentrum Berlin, Berlin, Germany